CLINICAL TRIAL: NCT06940063
Title: Does Active Music-Based Intervention Alter Cognitive Function, Sensitivity to Stimuli, Pain Catastrophizing and Quality of Life in Patients With Chronic Low Back Pain?
Brief Title: Active Music-Based Intervention in Patients With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sharon Wang-Price (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Sponsor-Investigator, Sharon Wang-Price, Professor/Faculty, Texas Woman's University
Organization: Texas Woman's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2025-89
Record Dates: First submitted 2025-04-02; First posted 2025-04-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain
Keywords: Music therapy; Central sensitization; chronic low back pain; cognitive function

STUDY DESIGN:
Intervention Model Description: Clinical trial with a single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active music-based in tervention (Experimental): Active musical interventions include playing an instrument, singing, or songwriting.
  Interventions: Procedure: Active music-based intervention

INTERVENTIONS:
Procedure: Active music-based intervention — Musical experience includes playing an instrument, singing, or songwriting.

SUMMARY:
The goal of this clinical trial is to learn if active music-based intervention works to treat patients with chronic low back pain. The main questions it aims to answer are:

1. Does active music-based intervention improve cognitive function?
2. Does active music -based intervention improve sensitivity to stimuli?
3. Does active music-based intervention improve pain catastrophizing behavior?
4. Does active music-based intervention improve quality of life?

Participant will visit the clinic for 5 sessions of assessments and active music-based intervention over 2 weeks. On the first visit, it will take each participant 45 minutes to complete the pre-intervention assessments followed by a 45-minute active music-based intervention. The active music-based intervention will last about an hour for the remaining 4 visits. On the 5th or last visit, after the one-hour intervention, it will take another 30 minutes for each participant to complete the post-intervention assessments.

DETAILED DESCRIPTION:
A prospective pre- and post-test research design will be used to compare outcome measures before and after the active music-based intervention (MBI) for the primary purpose of this study: to examine the effects of active MBI on cognitive function, sensitivity to stimuli, pain catastrophizing behavior and quality of life in individuals with chronic low back pain (CLBP). The secondary purpose of the study is to determine if there is a difference in cognitive function between participants with high vs. low levels of central sensitization, and to examine whether active music-based intervention (MBI) has differential effects on cognitive function and sensitivity to pressure stimuli.

After the eligible participants are enrolled in the study, each participant will be asked to complete an intake form to collect their demographic data (e.g., age, sex, race, height, weight, and occupation), past medical history, and questions related to their low back pain (onset, injury mechanism if any, location, duration, type, and nature). In addition, pain intensity and disability level will be determined using the Numerical Pain Rating Scale (NPRS) and the Modified Oswestry Low Back Pain Disability Questionnaire (OSW), respectively. The data collected will be used to describe the participants' characteristics of the study sample. Lastly, the severity of central sensitization will be determined by the Central Sensitization Inventory (CSI). A cutoff score of 33.5 from the CSI will be used to dichotomize the participants into the high vs. low level of CS. The target sample size is 40, 20 with a high level of central sensitization (CSI score of 33.5 or higher) and 20 with a low level of central sensitization (CSI score < 33.5).

Each participant will complete the outcome measurements before and after 5 sessions of active MBI. The primary outcome measures include cognitive tests, the pressure pain threshold (PPT) test, the Pain Catastrophizing Scale and the Patient-Reported Outcomes Measurement Information System - 29 (PROMIS-29) - see details in the Outcome Measure section.

There will be 5 intervention sessions. The first intervention will be administered after the outcome measure assessments and will last about 45 minutes. The other 4 intervention sessions will be one hour in length. During the first session, each participant will choose a preferred active musical experience in which they will engage for the entire study, including playing an instrument, singing, or songwriting. When the participants choose instrument playing or singing, they also will be given options to play a music piece or sing a song that they already know or that they can improvise. An example of improvisation is playing on a piano a piece of music which was written for violin.

All of the intervention sessions will be conducted by research assistants who are board-certified, credentialed music therapists. These researchers are trained in assessment, intervention planning, and treatment implementation. All of the intervention sessions will occur in a music therapy clinic at Texas Woman's University - Denton, Department of Music Therapy that is equipped with a wide variety of musical instruments, playback equipment, and ambient lighting.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-65 years of age
* have chronic low back pain (CLBP) primarily in the L4-5 area. The CLBP is defined as a back pain problem that has persisted at least 3 months and has resulted in pain on at least half the days in the past 6 months.

Exclusion Criteria:

Participants will be excluded if their low back pain (LBP) is due to a non-musculoskeletal origin or they have any medical conditions that may affect the results:

* Previous back surgery
* Systemic arthritis (e.g., rheumatoid arthritis, psoriatic arthritis).
* Fracture of thoracic and lumbar spine, pelvis
* Infection
* Tumor
* Traumatic brain injury
* Stroke
* Seizures/epilepsy
* Any other neurological disease (e.g., multiple sclerosis, muscular dystrophy, - Parkinson's)
* Circulation/vascular problems (e.g., Raynaud's)
* Cancer
* Uncontrolled diabetes/high blood sugar
* Currently pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | This outcome measure (SCWT) will be administered twice, before the start of treatment and after the end of treatment at 2 weeks.
  Cognitive function will be assessed using the Stroop Color and Word Test (SCWT).
  The SCWT is used to measure a person's attentional interference or the ability to inhibit the interference of a second stimulus while continuing to process an original stimulus. A computerized version of the SCWT via a software program DirectRT (Empirisoft Corp., New York, NY) will be used. The SCWT consists of 3 parts, each containing 24 consecutive stimuli. A reaction time will be computed in software based on the speed of the participant's response.
Cognitive function | This outcome measure (CTMT2) will be administered twice, before the start of treatment and after the end of treatment at 2 weeks.
  Cognitive function will be assessed using the Comprehensive Trail Making Test - Second Edition (CTMT2).
  The CTMT2 consists of 5 trails requiring cognitive control between competing stimuli and schemas. Trails 1-3 measure inhibitory control by completing trails with increasing numbers of distractors. Trails 4-5 measure set-shifting by requiring participants to shift between opposing mental sets (i.e., numbers and letters). The test will use standardized instructions.

SECONDARY OUTCOMES:
Sensitivity to stimuli | This outcome measure (PPT) will be administered twice, before the start of treatment and after the end of treatment at 2 weeks.
  Pressure pain threshold (PPT) will be used to determine the level of sensitivity to stimuli using a hand-held computerized pressure algometer (Medoc ltd., Ramat Yishai, Israel). The algometer will be pressed vertically on the most tender point of the participant's low back. To provoke the participant's pain or discomfort, pressure will be increased at a rate of 40 kPa/sec until the participant feels pain as indicated by pressing the patient safety button. Three trials of PPT testing will be administered.
Pain catastrophizing | This outcome measure (PCS) will be administered twice, before the start of treatment and after the end of treatment at 2 weeks.
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS). The PCS is a 13-item questionnaire that requires the participants to select their level of agreement for each item on a 5-point Likert scale. The total score ranges from 0-52, with a higher score indicating greater levels of pain catastrophizing
Health-related Quality of life | This outcome measure (PROMIS-29) will be administered twice, before the start of treatment and after the end of treatment at 2 weeks.
  Health-related quality of life will be determined by the Patient-Reported Outcomes Measurement Information System -29 (PROMIS-29). The PROMIS-29 is a 29-item questionnaire that assesses general health-related quality of life across 7 domains (i.e., physical function, pain interference, anxiety, depression, fatigue, sleep disturbance, and social roles) and pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wang-Price, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Department of Music, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Sharing IPD raises ethical concerns about participant privacy and the potential for misuse of sensitivity data. Data protection laws and regulations can restrict the sharing of personal data, even for research purposes.